CLINICAL TRIAL: NCT04327739
Title: Effects of Adding Two Different Types of Manual Techniques to a Therapeutic Exercise Program for the Management of Chronic Neck Pain: A Randomized Controlled Trial of Comparative Effectiveness
Brief Title: Adding Two Different Types of Manual Techniques to an Exercise Program for the Management of Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, LYTRAS DIMITRIOS, Dimitrios Lytras PT, Phd, Postdoctoral Research Fellow, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 256445/2019
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Neck Pain
Keywords: Chronic Neck Pain; Exercise; Manual techniques; Spinal manipulation; Integrated neuromuscular inhibition technique; Rehabilitation
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: An assessor-blind randomized control trial with a duration of ten weeks and a 6-month follow up will be performed in 80 women with chronic neck pain. The participants will be allocated into four groups of 20 persons each (three intervention groups and one control group). The first three groups will follow the same exercise program. Only exercise will be applied to the first group. The second group will apply a combination of soft tissue mobilization techniques and exercise. The third group will follow a combination of spinal manipulation and exercise, while the fourth group will not receive any treatment
Who Masked: Outcomes Assessor
Masking Description: Assessor-blind randomized control trial. A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1 Exercise (Experimental): Participants allocated to this group received a 10 weeks exercise programme for neck and upper limbs muscles
  Interventions: Other: Intervention 1 Exercise
- Intervention 2 Exercise and INIT (Experimental): Participants allocated to this group received the same exercise programme as group 1 in combination with the integrated neuromuscular inhibition technique (INIT)
  Interventions: Other: Intervention 2 Exercise and INIT
- Intervention 3 Exercise and SMT (Experimental): Participants allocated to this group received the same exercise programme as group 1 in combination with cervical manipulation
  Interventions: Other: Intervention 3 Exercise and SMT
- Control (Placebo Comparator): Participants allocated to this group received general consulting instructions and a home based general exercise sheet
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention 1 Exercise — • Exercise programme Endurance and Resistant training exercise program (Duration: 45 minutes) • Muscle retraining of longus colli and endurance training of the deep cervical flexors. • Resistant exercises for the muscles involved in neck flexion, extension, side bending and rotation of the neck region. Isometric contractions exercises (20-70% of MVC) and resistant exercises (12-15RM). • Active ROM exercises for the neck muscles • Upper limbs exercises with resistant bands • Stretching exercises for the neck and upper limbs muscles
  Arms: Intervention 1 Exercise
Other: Intervention 2 Exercise and INIT — * Exercise programme same as Intervention Group 1 and
  * Integrated Neuromuscular Inhibition Technique application. Integrated Neuromuscular Inhibition Technique application. (Duration: 15min) The protocol was applied to the following muscles: • Upper border of the trapezius muscle • sternocleidomastoid • levator scapulae muscle • splenius capitis muscle Integrated Neuromuscular Inhibition Technique includes the combination of the following technique: • Ischemic compression • Muscle energy technique • Straincounterstrain technique
  Arms: Intervention 2 Exercise and INIT
Other: Intervention 3 Exercise and SMT — * Exercise programme same as Intervention Group 1 and
  * Manipulation Care. Participants allocated to this group received Spinal Manipulation Therapy after the therapeutic exercise programme. Treatment was delivered by 1 chiropractor with a minimum 5-year experience of clinical practice. Pain provocation and static/motion palpation findings were used to determine areas of treatment in the cervical spine. The Manipulation Therapy technique included joint motion using a diversified thrust technique, and mobilization, a low-velocity type of joint oscillation. The type and the force of the applied spinal manipulation were individualized according to the age and physical condition of each participant. Soft passive stretching, light massage and hot packs were applied to the cervical and upper thoracic area before manipulation in order to prepare each participant.
  Arms: Intervention 3 Exercise and SMT
Other: Control — Participants allocated to this group received general consulting istructions and a home based general exercise sheet
  Arms: Control

SUMMARY:
Neck pain is one of the most common and costly musculoskeletal disorders in western societies with a high rate of recurrence and chronicity. In chronic neck pain, the persistence of symptoms is highly associated with changes in the biomechanics of the neck region that are related to the muscular imbalance between the neck muscles and specifically between the deep and superficial neck flexors. Manual techniques are special techniques applied by hand from the therapist that focus on reducing symptoms and improving disability. Both spinal manipulation and soft tissue mobilization techniques have a positive effect in individuals with chronic neck pain, especially when they are combined with the appropriate therapeutic exercise programme. However, it has not been determined which of the above-mentioned combinations is more effective in patients with chronic neck pain.

The aim of this study is to compare the efficacy of two different kinds of manual technique, when they combine with the same therapeutic exercise program in the management of patients with chronic neck pain.

An assessor-blind randomized control trial with a duration of ten weeks and a 6-month follow up will be performed in 80 women with chronic neck pain. The participants will be allocated into four groups of 20 persons each (three intervention groups and one control group). The first three groups will follow the same exercise program. Only exercise will be applied to the first group. The second group will apply a combination of soft tissue mobilization techniques and exercise. The third group will follow a combination of spinal manipulation and exercise, while the fourth group will not receive any treatment. The neck pain will be evaluated with the visual analogue scale, the disability related to neck pain with the neck disability index, the pressure pain threshold of the neck muscles with pressure algometry, the active range of motion with a bubble inclinometer, the maximum isometric strength of the neck muscles with a hand dynamometer, the muscular fatigue of the flexors of the neck with the craniocervical flexion test and the quality of life with the sf-36 questionnaire before, during and after the intervention, while follow-ups will take place six months later.

DETAILED DESCRIPTION:
Background Neck pain is one of the most common and costly musculoskeletal disorders in western societies with a high rate of recurrence and chronicity. In chronic neck pain, the persistence of symptoms is highly associated with changes in the biomechanics of the neck region that are related to the muscular imbalance between the neck muscles and specifically between the deep and superficial neck flexors. Manual techniques are special techniques applied by hand from the therapist that focus on reducing symptoms and improving disability. Both spinal manipulation and soft tissue mobilization techniques have a positive effect in individuals with chronic neck pain, especially when they are combined with the appropriate therapeutic exercise programme. However, it has not been determined which of the above-mentioned combinations is more effective in patients with chronic neck pain.

Aim The aim of this study is to compare the efficacy of two different kinds of manual technique, when they combine with the same therapeutic exercise program in the management of patients with chronic neck pain.

Method An assessor-blind randomized control trial with a duration of ten weeks and a 6-month follow up will be performed in 80 women with chronic neck pain. The participants will be allocated into four groups of 20 persons each (three intervention groups and one control group). The first three groups will follow the same exercise program. Only exercise will be applied to the first group. The second group will apply a combination of soft tissue mobilization techniques and exercise. The third group will follow a combination of spinal manipulation and exercise, while the fourth group will not receive any treatment. The neck pain will be evaluated with the visual analogue scale, the disability related to neck pain with the neck disability index, the pressure pain threshold of the neck muscles with pressure algometry, the active range of motion with a bubble inclinometer, the maximum isometric strength of the neck muscles with a hand dynamometer, the muscular fatigue of the flexors of the neck with the craniocervical flexion test and the quality of life with the sf-36 questionnaire before, during and after the intervention, while follow-ups will take place six months later.

ELIGIBILITY:
Inclusion Criteria:

* Women with chronic neck pain with a duration of symptoms for at least three months
* Existence of at least one active or latent trigger point in any of the muscles: levator scapulae, upper trapezoid, and splenius capitis
* Patients whose neck pain has emerged as a result of a specific pathology, confirmed by radio-diagnostic tests (X-ray or MRI)
* Patients with a medical referral for physical therapy with the etiology of neck pain

Exclusion Criteria:

* Included the acute stage of symptoms confirmed by visual analog scale (VAS; score >70 mm)
* Participation in any kind of treatment during the past 3 months (e.g., physiotherapy, massage, local injections of anesthetic blocks)
* Participation in an exercise program concerning the neck muscles during the past 6 months
* Background of neck trauma and/or surgery in the neck region
* Inflammatory muscle diseases, joint infections, and malignancy.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with visual analogue scale (VAS) | pre-treatment, Week: 2, 4, 6,10, 34
  VAS is a card with an uncalibrated scale ranging from 0-100 mm on the one side (with zero representing no pain and 100 representing the worst pain in life) with each millimeter representing one pain level. The patient subjectively estimated his or her pain level by marking a vertical line on the uncalibrated scale between zero and one hundred. Then the exact value of pain intensity could be obtained with a single ruler. Hence, the higher the value, the more intense the pain. VAS is widely used as it is easy to implement and is characterized by good psychometric properties.
Changes in Pressure Pain threshold with pressure algometry | pre-treatment, Week: 2, 4, 6, 10, 34
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT was assessed by a digital algometer. Pressure pain threshold was assessed over the upper border of the trapezius muscle halfway between the midline and the lateral border of the acromion, the levator scapulae muscle 2 cm above the lower insertion located in the upper medial border of the scapulae, Sternocleidomastoid muscle and to splenius capitis 2 cm lateral to the spinous processus of the axis. The metal rod of the algometer was placed vertically on the site and the examiner applied gradually increasing pressure at a rate of 1Kg/s. PPT was calculated in kg/cm2.
Changes in functional capacity with the Greek Version of Neck disability index questionnaire | pre-treatment, Week 6, 10, 34
  It is a self-reported ten-item scale. Each item assesses different neck pain complaints. Most of the items are related to restrictions in activities of daily living, and each item is expressed by 6 different assertions in the range 0-5, with 0 indicating no disability and 5 indicating the highest disability. The total score ranges from 0 to 50. Disability Index (NDI) has sufficient support in the literature, being the most commonly used to report neck pain.
Changes in maximum isometric strength of neck muscles with Manual Muscular Testing | pre-treatment, Week: 2, 4, 6, 10, 34
  Cervical flexion, extension, and side bending isometric strength were assessed using a Manual Muscular Testing device with the participants in supine and prone position. Isometric strength were assessed in kg.
Changes in Cervical Range of Motion with bubble inclinometers | pre-treatment, Week: 2, 4, 6, 10, 34
  Cervical active range of motion was measured with 2 bubble inclinometers. One was placed on the top of the head and the second on the spinous process of C7.Active cervical flexion, extension and side bending range of motion were assessed with participants sitting in upright position. Range of motion was measured in degrees
Changes in deep flexors muscle endurance with craniocervical flexion test | pre-treatment, Week: 2, 4, 6, 10, 34
  The craniocervical flexion test (CCFT) is a clinical test of the anatomical action of the deep cervical flexor muscles, (longus capitis, and longus colli). It could be described as a test of neuromotor control. It includes the performance of five progressive stages of increasing craniocervical flexion range of motion (22, 24, 26, 28, and 30 mm Hg). It is a low-load test performed in the supine position with the patient guided to each stage by feedback from a pressure sensor placed behind the neck. While the test in the clinical setting provides only an indirect measure of performance.
Changes in quality of life with the sort form of SF-36 Health Survey | pre-treatment, Week: 10, 34
  For the evaluation of the intervention in the quality of life of the participants the short form of SF-36 Health Survey questionnaire was used. SF-36 consists of 36 questions, selected from the Medical Outcomes Study (MOS), which relate to eight different parameters of mental and physical health. Total Physical and Mental Health, as well as the subcategory of Bodily Pain were evaluated in this study

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Sykaras, PT, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (2):
- Greece (2):
  - Aristotle University of Thessaloniki, Thessaloniki, Central Makedonia
  - Department of Physical Education and Sports Sciences, Thessaloniki, Thermi

IPD SHARING:
Plan to Share IPD: No